CLINICAL TRIAL: NCT01123122
Title: A Comparison of Strict Glucose Control With Usual Care at the Time of Islet Cell Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Vancouver Coastal Health (Other Government)
Responsible Party: David M. Thompson, Vancouver General Hospital Department of Endocrinology and Metabolism
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHEndo0510
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus, Type 1; Islet Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strict glucose control (Active Comparator)
  Interventions: Other: Strict glucose control
- Standard glucose control (No Intervention)

INTERVENTIONS:
Other: Strict glucose control — Blood glucose level to be maintained at 4-6 mmol/L at the time of islet transplantation until two weeks post-transplantation.
  Arms: Strict glucose control

SUMMARY:
Islet transplants for those with type 1 diabetes have enabled many to initially eliminate insulin, however, only a fraction of the transplanted cells typically survive and the functioning of these decrease over time. As a result, most patients will eventually require some insulin. Currently, the cause of this poor survival and decrease in function is not understood; although previous research has demonstrated that even a slightly elevated level of blood glucose can impair islet function. This study will determine if strict blood glucose control at the time of islet transplantation, when the cells are the most fragile, will improve the survival and functioning of transplanted islet cells three months after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* more than 5 years since diagnosis of diabetes
* c-peptide negative

Exclusion Criteria:

* ischemic heart disease
* previous transplant
* recurrent infections
* malignancy (except basal or squamous skin cancer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Islet cell function | Three months
  Function will be assessed three months post-transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: David M Thompson, MD, Principal Investigator — Vancouver General Hospital Department of Endocrinology and Metabolism
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004
- [Background] Shapiro AM, Ricordi C, Hering B. Edmonton's islet success has indeed been replicated elsewhere. Lancet. 2003 Oct 11;362(9391):1242. doi: 10.1016/S0140-6736(03)14526-6. No abstract available. PMID 14568760
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207
- [Background] Rickels MR, Schutta MH, Markmann JF, Barker CF, Naji A, Teff KL. beta-Cell function following human islet transplantation for type 1 diabetes. Diabetes. 2005 Jan;54(1):100-6. doi: 10.2337/diabetes.54.1.100. PMID 15616016
- [Background] Eich T, Eriksson O, Lundgren T; Nordic Network for Clinical Islet Transplantation. Visualization of early engraftment in clinical islet transplantation by positron-emission tomography. N Engl J Med. 2007 Jun 28;356(26):2754-5. doi: 10.1056/NEJMc070201. No abstract available. PMID 17596618
- [Background] Froud T, Ricordi C, Baidal DA, Hafiz MM, Ponte G, Cure P, Pileggi A, Poggioli R, Ichii H, Khan A, Ferreira JV, Pugliese A, Esquenazi VV, Kenyon NS, Alejandro R. Islet transplantation in type 1 diabetes mellitus using cultured islets and steroid-free immunosuppression: Miami experience. Am J Transplant. 2005 Aug;5(8):2037-46. doi: 10.1111/j.1600-6143.2005.00957.x. PMID 15996257
- [Background] Pfeifer MA, Halter JB, Porte D Jr. Insulin secretion in diabetes mellitus. Am J Med. 1981 Mar;70(3):579-88. doi: 10.1016/0002-9343(81)90579-9. PMID 7011013
- [Background] Brunzell JD, Robertson RP, Lerner RL, Hazzard WR, Ensinck JW, Bierman EL, Porte D Jr. Relationships between fasting plasma glucose levels and insulin secretion during intravenous glucose tolerance tests. J Clin Endocrinol Metab. 1976 Feb;42(2):222-9. doi: 10.1210/jcem-42-2-222. PMID 1262429
- [Background] Godsland IF, Jeffs JAR, Johnston DG. Loss of beta cell function as fasting glucose increases in the non-diabetic range. Diabetologia. 2004 Jul;47(7):1157-1166. doi: 10.1007/s00125-004-1454-z. Epub 2004 Jul 13. PMID 15249997
- [Background] Moran A, Zhang HJ, Olson LK, Harmon JS, Poitout V, Robertson RP. Differentiation of glucose toxicity from beta cell exhaustion during the evolution of defective insulin gene expression in the pancreatic islet cell line, HIT-T15. J Clin Invest. 1997 Feb 1;99(3):534-9. doi: 10.1172/JCI119190. PMID 9022089
- [Background] Donath MY, Gross DJ, Cerasi E, Kaiser N. Hyperglycemia-induced beta-cell apoptosis in pancreatic islets of Psammomys obesus during development of diabetes. Diabetes. 1999 Apr;48(4):738-44. doi: 10.2337/diabetes.48.4.738. PMID 10102689
- [Background] Pick A, Clark J, Kubstrup C, Levisetti M, Pugh W, Bonner-Weir S, Polonsky KS. Role of apoptosis in failure of beta-cell mass compensation for insulin resistance and beta-cell defects in the male Zucker diabetic fatty rat. Diabetes. 1998 Mar;47(3):358-64. doi: 10.2337/diabetes.47.3.358. PMID 9519740
- [Background] El-Assaad W, Buteau J, Peyot ML, Nolan C, Roduit R, Hardy S, Joly E, Dbaibo G, Rosenberg L, Prentki M. Saturated fatty acids synergize with elevated glucose to cause pancreatic beta-cell death. Endocrinology. 2003 Sep;144(9):4154-63. doi: 10.1210/en.2003-0410. PMID 12933690
- [Background] Boden G, Chen X. Effects of fat on glucose uptake and utilization in patients with non-insulin-dependent diabetes. J Clin Invest. 1995 Sep;96(3):1261-8. doi: 10.1172/JCI118160. PMID 7657800
- [Background] Boden G, Jadali F, White J, Liang Y, Mozzoli M, Chen X, Coleman E, Smith C. Effects of fat on insulin-stimulated carbohydrate metabolism in normal men. J Clin Invest. 1991 Sep;88(3):960-6. doi: 10.1172/JCI115399. PMID 1885781
- [Background] Roden M, Price TB, Perseghin G, Petersen KF, Rothman DL, Cline GW, Shulman GI. Mechanism of free fatty acid-induced insulin resistance in humans. J Clin Invest. 1996 Jun 15;97(12):2859-65. doi: 10.1172/JCI118742. PMID 8675698
- [Background] Maedler K, Spinas GA, Dyntar D, Moritz W, Kaiser N, Donath MY. Distinct effects of saturated and monounsaturated fatty acids on beta-cell turnover and function. Diabetes. 2001 Jan;50(1):69-76. doi: 10.2337/diabetes.50.1.69. PMID 11147797
- [Background] Cnop M, Hannaert JC, Hoorens A, Eizirik DL, Pipeleers DG. Inverse relationship between cytotoxicity of free fatty acids in pancreatic islet cells and cellular triglyceride accumulation. Diabetes. 2001 Aug;50(8):1771-7. doi: 10.2337/diabetes.50.8.1771. PMID 11473037
- [Background] Markmann JF, Deng S, Huang X, Desai NM, Velidedeoglu EH, Lui C, Frank A, Markmann E, Palanjian M, Brayman K, Wolf B, Bell E, Vitamaniuk M, Doliba N, Matschinsky F, Barker CF, Naji A. Insulin independence following isolated islet transplantation and single islet infusions. Ann Surg. 2003 Jun;237(6):741-9; discussion 749-50. doi: 10.1097/01.SLA.0000072110.93780.52. PMID 12796569
- [Background] Warnock GL, Meloche RM, Thompson D, Shapiro RJ, Fung M, Ao Z, Ho S, He Z, Dai LJ, Young L, Blackburn L, Kozak S, Kim PT, Al-Adra D, Johnson JD, Liao YH, Elliott T, Verchere CB. Improved human pancreatic islet isolation for a prospective cohort study of islet transplantation vs best medical therapy in type 1 diabetes mellitus. Arch Surg. 2005 Aug;140(8):735-44. doi: 10.1001/archsurg.140.8.735. PMID 16103282
- [Background] Warnock GL, Thompson DM, Meloche RM, Shapiro RJ, Ao Z, Keown P, Johnson JD, Verchere CB, Partovi N, Begg IS, Fung M, Kozak SE, Tong SO, Alghofaili KM, Harris C. A multi-year analysis of islet transplantation compared with intensive medical therapy on progression of complications in type 1 diabetes. Transplantation. 2008 Dec 27;86(12):1762-6. doi: 10.1097/TP.0b013e318190b052. PMID 19104418
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] ADVANCE Collaborative Group; Patel A, MacMahon S, Chalmers J, Neal B, Billot L, Woodward M, Marre M, Cooper M, Glasziou P, Grobbee D, Hamet P, Harrap S, Heller S, Liu L, Mancia G, Mogensen CE, Pan C, Poulter N, Rodgers A, Williams B, Bompoint S, de Galan BE, Joshi R, Travert F. Intensive blood glucose control and vascular outcomes in patients with type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2560-72. doi: 10.1056/NEJMoa0802987. Epub 2008 Jun 6. PMID 18539916
- [Background] Krinsley JS. Effect of an intensive glucose management protocol on the mortality of critically ill adult patients. Mayo Clin Proc. 2004 Aug;79(8):992-1000. doi: 10.4065/79.8.992. PMID 15301325
- [Background] Rickels MR, Naji A, Teff KL. Acute insulin responses to glucose and arginine as predictors of beta-cell secretory capacity in human islet transplantation. Transplantation. 2007 Nov 27;84(10):1357-60. doi: 10.1097/01.tp.0000287595.16442.a7. PMID 18049122